CLINICAL TRIAL: NCT07095283
Title: Second-generation Radiofrequency Application and Specific Therapeutic Exercise as a Treatment for Stress Urinary Incontinence Due to Urethral Instability. Randomised Clinical Trial
Brief Title: Second-generation Radiofrequency Application and Therapeutic Exercise for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Clinical Professor, Cardenal Herrera University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CEEI25/646
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stress Urinary Incontinence
Keywords: urethral instability; radiofrequency; physical exercise; functional ultrasound; quality of life
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RF Therapy (Experimental): Participants will be placed in the lithotomy position. The treatment temperature will be set at 41°C, with a frequency of 1 MHz and power of 75 kJ. Once the indicated temperature has been reached, the physical therapist will perform small upward and downward movements along the urethral canal, dividing the time equally between both sides. One RF session will be performed every 7 days, as described by the author, for a total of 5 sessions. We divided the subjects into mild SUI (1-2 points in the Sandvik test); moderate SUI (Sandvik test of 3 to 6 points), severe SUI (8-9 points Sandvik test); and very severe SUI (12 points in Sandvik test).
  Interventions: Diagnostic Test: Short International Consultation on Incontinence Questionnaire (ICIQ-SF); Diagnostic Test: King's Health Questionnaire (KHQ); Diagnostic Test: Ultrasound evaluation; Diagnostic Test: Sandvik Severity Index; Diagnostic Test: Oxford's scale; Diagnostic Test: Biofeedback
- Pelvic floor muscle training (PFMT) (Experimental): The PFMT will consist of a targeted program with a protocol of core and pelvic floor exercises established based on an assessment of the patients' strength, endurance, and fatigue, with a frequency of twice a week led by a physical therapist and a duration of 45 minutes each day for a period of 16 weeks. It will be carried out in groups of 8 people and accompanied by a physical therapist experienced in therapeutic exercise. We divided the subjects into mild SUI (1-2 points in the Sandvik test); moderate SUI (Sandvik test of 3 to 6 points), severe SUI (8-9 points Sandvik test); and very severe SUI (12 points in Sandvik test).
  Interventions: Diagnostic Test: Short International Consultation on Incontinence Questionnaire (ICIQ-SF); Diagnostic Test: King's Health Questionnaire (KHQ); Diagnostic Test: Ultrasound evaluation; Diagnostic Test: Sandvik Severity Index; Diagnostic Test: Oxford's scale; Diagnostic Test: Biofeedback
- combination of RF Therapy and PFMT (Experimental): We divided the subjects into mild SUI (1-2 points in the Sandvik test); moderate SUI (Sandvik test of 3 to 6 points), severe SUI (8-9 points Sandvik test); and very severe SUI (12 points in Sandvik test).
  Interventions: Diagnostic Test: Short International Consultation on Incontinence Questionnaire (ICIQ-SF); Diagnostic Test: King's Health Questionnaire (KHQ); Diagnostic Test: Ultrasound evaluation; Diagnostic Test: Sandvik Severity Index; Diagnostic Test: Oxford's scale; Diagnostic Test: Biofeedback

INTERVENTIONS:
Diagnostic Test: Short International Consultation on Incontinence Questionnaire (ICIQ-SF) — This is a self-administered questionnaire with four questions and a total score ranging from 0 [best] to 21 [worst] that identifies people with urinary incontinence and its impact on quality of life.
Diagnostic Test: King's Health Questionnaire (KHQ) — The KHQ is a self-administered instrument specifically designed to assess quality of life in women with UI. It consists of 21 items distributed across 9 dimensions: perception of overall health (1 item), impact of UI (1 item), limitations in daily activities (2 items), physical limitations (2 items), social limitations (2 items), personal relationships (3 items), emotions (3 items), sleep/energy (2 items), and severity of UI (5 items). The score range for each dimension is from 0 (lowest impact of UI and therefore best quality of life) to 100 (highest impact, worst quality of life). This questionnaire provides an overall value for the quality of life of the patient with UI (Overall Score-OS) and another specific value for each dimension on a scale with the following range: 0: Best possible quality of life - 100: Worst possible quality of life.
Diagnostic Test: Ultrasound evaluation — A two-dimensional (2D) ultrasound system with B-mode capability and cine-loop function, a 3.5 to 6 MHz curved convex probe transducer, was used for the perineal image. The examination will be performed in the dorsal lithotomy position, with the hips flexed and slightly abducted and the heels placed close to the buttocks, or in a standing position if necessary.
Diagnostic Test: Sandvik Severity Index — It allows the severity of UI to be determined based on two questions. Interpretation based on the score is classified as follows: 1-2 mild UI, 3-6 moderate UI, 8-9 severe UI, 12 very severe UI.
Diagnostic Test: Oxford's scale — The strength of the Pelvic floor muscles will be evaluated digitally using functional ultrasound and classified according to the Oxford scale.
Diagnostic Test: Biofeedback — Muscular (mmHg) and static strength (seconds); Fatigability or Dynamic Endurance (% and cmH₂O)
  Other Names: Muscular and static strength; Fatigability or Dynamic Endurance

SUMMARY:
Stress urinary incontinence (SUI) is defined as the loss of the ability to hold urine after exertion, i.e., as a result of imbalances in intra-abdominal pressure, which directly affect the lower urinary tract. SUI has been shown to have a significant impact on the quality of life of those affected, impacting physical, social, and psycho-emotional aspects. Among the proposed treatments is a physiotherapeutic approach, which is offered as a less invasive and painless therapy with fewer adverse effects than pharmacological or surgical treatment. Pelvic floor muscle training (PFMT) is the most effective physiotherapeutic treatment for SUI, increasing the contractile capacity of the muscles and restoring stability throughout the pelvic diaphragm, thereby ensuring proper support of the pelvic organs. Radiofrequency (RF) therapy is currently being proposed as a therapeutic option that may offer certain advantages over those reported for photoplethysmography (PPMT). The potential benefits of RF therapy are attributed to its ability to stimulate collagen metabolism, thereby promoting tissue regeneration. Radiofrequency (RF) is a non-invasive and painless method that has the potential to yield analogous results to pelvic physical therapy (PPMT) as a standalone treatment or enhance the efficacy of PPMT when administered in conjunction with RF for stress urinary incontinence (SUI).

The objective of the present study is to analyse the effectiveness of PFMT and RF as single or combined treatments for SUI in women at Clínica Traña, a clinic specialising in the treatment of pelvic floor dysfunction in Costa Rica. Following the process of obtaining informed consent, patients will be offered a single or combined treatment of RF and/or PFMT. The strength of the pelvic floor muscles, pelvic function and the impact of pelvic dysfunctions on quality of life will be evaluated with a one-year follow-up after the conclusion of treatment.

The project possesses the facilities, equipment, and personnel necessary to ensure its viability, as well as proven clinical experience.

The scientific and technical impact of the proposed treatment protocol will be achieved by establishing an effective therapeutic strategy to address SUI. The social impact of SUI is significant, given its high prevalence and the fact that it has physical consequences as well as a negative impact on the social activities, work functions and emotions of women who suffer from it.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 who meet the International Continence Society (ICS)
* diagnostic criteria for SUI, which consists of involuntary leakage of urine during increased intra-abdominal pressure in the absence of bladder contractions such as coughing, sneezing, and other physical activities.

Exclusion Criteria:

* diagnosis of urgent or mixed UI
* diagnosis of pelvic organ prolapse
* taking any treatment for UI
* pregnancy
* history of pelvic surgery, urinary tract infection, or diagnosed psychological disorders
* presence of scars, malformations, abnormal pelvic masses, tissue irritation, or any other condition in the area that could be causing pelvic and urinary function problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire (ICIQ-SF) | Pre - post intervention; after 3,6,12 months
  0 to 21 points, where higher scores indicate greater impact of incontinence
King´s Health Questionnaire (KHQ) | Pre - post intervention; after 3,6,12 months
  0 to 100, where 0 indicates the best quality of life and 100 the worst
ultrasound analysis: Resting aperture (Ar) | Pre - post intervention; after 3,6,12 months
  degrees
ultrasound analysis: Opening during exertion (Ae) | Pre - post intervention; after 3,6,12 months
  degrees
Opening difference (Ae-Ar) | Pre - post intervention; after 3,6,12 months
  degrees
MUSCULAR STRENGTH | Pre - post intervention; after 3,6,12 months
  defined as the ability of tissue to generate tension based on its contractile capacity, being the best of three attempts to contract, assessed using the modified OXFORD scale
Function of the pelvic floor muscles | Pre - post intervention; after 3,6,12 months
  The best of the three attempts is selected, graded as follows: 0 = no contraction, 1 = partial contraction, 2 = contraction of the pelvic floor muscles + contraction of related muscles, 3 = isolated contraction of the Pelvic floor muscles
STATIC MUSCLE STRENGTH | Pre - post intervention; after 3,6,12 months
  the ability to maintain optimal contraction (isometric, tonic fibers) for as long as possible, measuring the seconds until fatigue sets in. ORDER: "contract and hold," taking the average of the three assessments.
Fatigability or Dynamic Endurance | Pre - post intervention; after 3,6,12 months
  maximum number of contractions in a unit of time, taking 10 seconds as the average. ORDER: "contract as many times as possible and at the highest speed," with the measurement being the average of the three assessments.
Oxford's Scale | Pre - post intervention; after 3,6,12 months
  allows the contractile capacity of the pelvic floor muscles to be assessed. It scores from 0 to 5, as follows: if there is no contraction, it is scored as 0; if the contraction is very weak, it is scored as 1; if the contraction is weak, it is scored as 2; if the contraction is moderate/with tension/and sustained, it is scored as 3; if the contraction is good and maintains tension with resistance, it is scored as 4; and if the contraction is strong and maintains tension against a resistant force, it is scored as 5.
Sandvik Severity Index | Pre - post intervention; after 3,6,12 months
  It allows the severity of UI to be determined based on two questions. Interpretation based on the score is classified as follows: 1-2 mild UI, 3-6 moderate UI, 8-9 severe UI, 12 very severe UI.

SECONDARY OUTCOMES:
age (years) | baseline
BMI (Body mass index) | baseline
  kg / m²
smoke | baseline
  yes/no
alcohol consumption | baseline
  yes/no
drug use | baseline
  yes/no
full-term pregnancies | baseline
  Number
natural childbirth | baseline
  yes/no
cesarean sections | baseline
  yes/no
tear | baseline
  yes/no
abortion | baseline
  yes/no
episiotomy | baseline
  yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- Ceu Cardenal Herrera University, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data associated with this paper will be available in the Zenodo repository
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2026-01-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT07095283/Prot_SAP_ICF_001.pdf